CLINICAL TRIAL: NCT02535832
Title: Skeletal Muscle Dysfunction in Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Beatriz Hanaoka, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0585-F6A
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis; Insulin Resistance
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): From the total participants enrolled into the cross-sectional study, the investigator will identify up to 18 participants who have insulin resistance and recruit them to participate in the placebo arm. Participants will take matching placebo throughout the 15 weeks of treatment.
  Interventions: Drug: Placebo
- Pioglitazone (Active Comparator): From the total participants enrolled into the cross-sectional study, the investigator will identify up to 18 participants who have insulin resistance and recruit them to participate in the pioglitazone arm. Participants will start by taking increasing doses for three weeks as follows: 1 capsule (15 mg) per day for 7 days, 1 capsule per day (30 mg) for 7 days, and 1 capsule (45mg), if tolerated. Participants will continue this dose (45 mg) throughout the 12 weeks of treatment.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone CT Scan DXA scan Needle muscle biopsy
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — Placebo CT Scan DXA scan Needle muscle biopsy
  Arms: Placebo

SUMMARY:
Muscle strength helps determine a person's quality of life and functional independence. Patients with rheumatoid arthritis often suffer from muscle weakness and a pre-diabetic condition called insulin resistance.

By doing this study, the investigators hope to learn why patients with rheumatoid arthritis (RA) suffer from muscle weakness.

DETAILED DESCRIPTION:
The investigator plans to enroll 80 participants with RA and 30 non-RA controls between the ages of 35 and 65 between August 2015 and December 2018 (arm-1). The investigator plan to perform a needle muscle biopsy in a subset of participants who agree to undergo this procedure. From the total cohort number of enrolled participants, 36 participants will be identified as having insulin resistance and recruit them to participate in the pioglitazone study (arm-2). Those patients who elect to participate further in the pioglitazone/ placebo study will sign separate consent document during Visit 1.

Since RA is more common in women, it is anticipated that 2/3 of the participants will be women. Children, pregnant or breast-feeding women, adults with impaired consent capacity, or vulnerable populations will not be enrolled.

In the cross-sectional study, after having provided informed consent, participants will undergo a history and physical exam by a rheumatologist to verify diagnosis of RA or that they are a healthy volunteer. All inclusion and exclusion criteria will be verified by the examining physician. During this visit, the participants will complete questionnaires including the Brief Pain Inventory (BPI), Health Assessment Questionnaire (HAQ), Patient Reported Outcomes Measurement Information System (PROMIS) questionnaire and SF-36. Participants will undergo dual energy x-ray absorptiometry (DXA) scanning to assess muscle mass of the upper leg (dominant and non-dominant sides), as well as computed tomography (CT) to assess body composition. Women of child bearing age will undergo urine pregnancy testing. Participants will undergo strength testing and a fatiguing bout of knee extension exercise. Blood will be drawn for glucose, insulin, liver function tests (LFT), lipid profile, rheumatoid factor (RF), anti-citrullinated protein antibodies (ACPA), insulin like growth factor (IGF-1), C-Reactive Protein (CRP), insulin like growth factor binding protein-1 (IGFBP-1) and insulin like growth factor binding protein-3 (IGFBP-3). All participants will be asked to wear an accelerometer for 7 day to measure physical activity. The participants will be scheduled to return to Center for Clinical and Translational Science (CCTS) within 7 days for biopsy of the vastus lateralis muscle.

In the pioglitazone clinical trial study, 36 participants who have insulin resistance will be recruited to receive pioglitazone. After the participants have provided informed consent, women of childbearing potential will be given a urine pregnancy test at visits 1, 3 and 6. The investigator will review participant eligibility and participants will be randomized to receive either pioglitazone 45 mg daily or matching placebo for 15 weeks. Below is the dosing schedule.

Participants will start by taking increasing doses for three weeks as follows: 1 capsule (15mg) per day for 7 days, 1 capsule per day (30 mg) for 7 days, and 1 capsule (45mg), if tolerated. Participants will continue this dose (45 mg) throughout the 10 weeks of treatment. The placebo or non-pioglitazone capsules will look identical to the pioglitazone capsules, but will contain inert substances, and the escalating dose schedule will be the same.

If participants experience difficulty with the drug, the investigators will slow the pace of dose escalation. If they cannot take 45 mg/day, then they may be dropped from the study. The placebo capsules will look identical to the pioglitazone capsules, but will contain inert substances. Drug compounding and dispensing (including blinding) will be handled by the University of Kentucky's Investigational Drug Service, which routinely serves this function. All participants in the pioglitazone study will undergo a second round of assessments. During the 15-week drug trial, participants will receive monthly phone calls to monitor for adverse effects. Additionally, participants will be asked to fill out a daily medication diary to monitor compliance and adverse effects. A skeletal muscle biopsy will be performed after treatment with pioglitazone/ placebo, which will take place within 1-2 weeks after the second round of assessments following pioglitazone treatment.

ELIGIBILITY:
Inclusion Criteria for RA patients (cross-sectional study):

* Age 35-65
* Diagnosed with RA by a Rheumatologist and according to American College of Rheumatology 2010 criteria

Inclusion Criteria for controls (cross-sectional study):

* Age 35-65
* In generally good health

Inclusion Criteria for RA patients who are: (i) insulin resistant by the 2-hour glucose tolerance test; (ii) have the presence of 3 or more risk factors for metabolic syndrome (MetS) according to the ATP III Clinical Identification of MetS criteria; (iii) have a Hemoglobin A1c level equal or greater than 5.7 and less than 6.5.

* Age 35-65
* Diagnosed with RA by a Rheumatologist and according to American College of Rheumatology 2010 criteria
* Insulin resistant according to the Matsuda index

Exclusion Criteria (cross-sectional study):

* Age <35 or >65
* Pregnant, breast-feeding, cognitive dysfunction, incarcerated or otherwise vulnerable persons
* Any acute or chronic medical or psychiatric disorder that, in the opinion of the investigators, would impair evaluation of the study measures

Exclusion criteria (pioglitazone randomized clinical trial):

* Women of reproductive age who are pregnant or who do not agree to effective birth control or who are lactating
* Clinically significant hepatic, cardiac or renal impairment
* Untreated osteoporosis
* Active cancer other than skin cancer
* Use of drugs (other than glucocorticoids) or nutritional supplements known to affect skeletal muscle mass
* Participation in regular and intense physical training
* Severe edema.

Exclusion criteria for the muscle biopsy (cross-sectional and pioglitazone randomized clinical trial):

* Bleeding diathesis or chronic anticoagulant therapy
* Unable or unwilling to discontinue aspirin or non-steroidal anti-inflammatory drugs for 5 days prior to muscle biopsy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Baseline
  2 hour oral glucose tolerance test will be performed after a 12-hour fast using 75 g glucose
Skeletal muscle strength in the quadriceps muscle | Changes from baseline and 12 weeks
  isometric strength test of the lower-extremity muscles (with one leg extension) using a Biodex to measure maximum voluntary isometric contraction (MVIC)
Monocytosis in peripheral blood | Changes from baseline and 12 weeks
  White blood cell populations will be isolated using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Hanaoka, MD MPH, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided